CLINICAL TRIAL: NCT03452462
Title: Electrical Resynchronization and Acute Hemodynamic Effects of Direct His Bundle Pacing Compared to Biventricular Pacing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Swiss National Fund for Scientific Research (Other)
Responsible Party: Principal Investigator, Haran Burri, MD, Professor, University Hospital, Geneva
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HisCRT_GVA
Record Dates: First submitted 2018-02-25; First posted 2018-03-02 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Cardiac Pacing, Artificial; Cardiac Resynchronization Therapy; Direct His Bundle Pacing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct His Bundle Pacing (Experimental): Pacing from the His bundle lead
  Interventions: Device: Pacing
- Biventricular Pacing (Active Comparator): Pacing from the right ventricular and coronary sinus leads
  Interventions: Device: Pacing

INTERVENTIONS:
Device: Pacing — Programming of either Direct His Bundle pacing or biventricular pacing

SUMMARY:
The aims are to compare Direct His Bundle Pacing (DHBP) with biventricular pacing (BiV) in terms of electrical resynchronization using electrocardiographic imaging (ECGI) and also in terms of acute hemodynamical effect using finger plethysmography and conduction velocimetry. The study will be a randomized crossover design with acute measurements.

DETAILED DESCRIPTION:
By recruiting native conducting tissue to relay electrical activation of the ventricles via the Purkinje fibre network, DHBP may potentially achieve greater electrical resynchronization and hemodynamic benefit compared to BiV where the electrical activation wavefronts propagate from two discrete pacing sites. Electrical synchrony achieved by these pacing modes have however never been compared. Furthermore, the acute hemodynamic effect of DHBP has been compared to BiV only in a small single study to date. The aims are to compare DHBP with BiV in terms of electrical resynchronization using electrocardiographic imaging (ECGI) and also in terms of acute hemodynamical effect using finger plethysmography and conduction velocimetry. The primary endpoint will be left ventricular activation time, with secondary endpoints including various electrical (right ventricular activation time, total ventricular activation time etc) and hemodynamic parameters (systolic pressure, cardiac output, cardiac contractility). It is expected that DHBP offers shorter left ventricular activation time (i.e. better synchrony) and hemodynamic benefit compared to BiV.

ELIGIBILITY:
Inclusion Criteria:

* Treatment of heart failure with a standard indication for CRT (NYHA III-IV, LVEF < 35% and QRS > 130ms; or LVEF< 40% and requirement for frequent ventricular pacing, irrespective of baseline QRS duration) and optimal medical treatment.

  * Permanent atrial fibrillation (allowing connection of the DHBP lead to the atrial port).
  * Patients implanted with 1) a CRT pacemaker or CRT defibrillator 2) a His lead with selective or non-selective DHBP, connected to the atrial port of the generator 3) a functional right ventricular lead and 4) a functional coronary sinus lead.
  * DHBP with selective or non-selective His capture

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Inability to undergo CT or an MRI (e.g. due to severe claustrophobia)
* Inability or refusal to sign the patient informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
Left ventricular activation time | 5 minutes
  Duration of left ventricular electrical activation

SECONDARY OUTCOMES:
Right ventricular activation time | 5 minutes
  Duration of right ventricular electrical activation
Total ventricular activation time | 5 minutes
  Duration of total ventricular electrical activation
Systolic pressure | 5 minutes
  Systolic blood pressure measured by finger plethysmography
Cardiac output | 5 minutes
  Cardiac output measured by conductive velocimetry
Cardiac contractility | 5 minutes
  Cardiac contractilit measured by conductive velocimetry

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zweerink A, Zubarev S, Bakelants E, Potyagaylo D, Stettler C, Chmelevsky M, Lozeron ED, Hachulla AL, Vallee JP, Burri H. His-Optimized Cardiac Resynchronization Therapy With Ventricular Fusion Pacing for Electrical Resynchronization in Heart Failure. JACC Clin Electrophysiol. 2021 Jul;7(7):881-892. doi: 10.1016/j.jacep.2020.11.029. Epub 2021 Feb 24. PMID 33640346